CLINICAL TRIAL: NCT03423446
Title: A Phase 1, Open-label, Parallel-group Study to Evaluate the Single-dose Pharmacokinetics of Telotristat Ethyl in Male and Female Subjects With Severe Hepatic Impairment and Matched Subjects With Normal Hepatic Function
Brief Title: Study to Evaluate the Pharmacokinetics of Telotristat Ethyl in Subjects With Severe Hepatic Impairment
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Lexicon Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LX1606.1-111-HEP; LX1606.111 (Other: Lexicon Pharmaceuticals, Inc.)
Record Dates: First submitted 2017-10-24; First posted 2018-02-06 (Actual); Last update posted 2018-10-15 (Actual); Status verified 2018-10

CONDITIONS: Hepatic Impairment
MeSH Terms: interventions — telotristat ethyl; telotristat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Severe Hepatic Impairment (Experimental): Up to 8 subjects with severe hepatic impairment (Child-Pugh Class C, score of 10 to 15 points)
  Interventions: Drug: Telotristat Ethyl
- Healthy Control (Experimental): Up to 8 healthy control subjects with normal hepatic function
  Interventions: Drug: Telotristat Ethyl

INTERVENTIONS:
Drug: Telotristat Ethyl — Telotristat ethyl (TE) 250 mg (1 x 250-mg tablet), single dose
  Other Names: telotristat etiprate, Xermelo

SUMMARY:
This study is designed to evaluate the effect of severe hepatic impairment on the pharmacokinetics (PK) of telotristat ethyl (TE) ( LP-778902 active moiety, metabolite), following administration of a single dose of TE 250 mg (1 x 250-mg tablet) compared to healthy, demographically-matched subjects with normal hepatic function.

ELIGIBILITY:
Inclusion Criteria:

* Adult male and female subjects ≥18 to ≤70 years of age, inclusive, at the time of Screening:

  1. Females of non-childbearing potential are to be surgically sterile (documented hysterectomy, tubal ligation, or bilateral salpingo-oophorectomy) or postmenopausal (defined as at least 12 months of spontaneous amenorrhea). Females of childbearing potential must agree to use an adequate method of contraception during the study from clinical research unit (CRU) admission through Safety Follow-up.

     Adequate methods of contraception for subjects or partner include condom, diaphragm, or cervical cap used in conjunction with spermicidal gel, foam, cream, film, or suppository. Hormonal contraception is NOT acceptable in this study. If necessary, follicle-stimulating hormone (FSH) results >40 IU/L at Screening are confirmatory in the absence of a clear postmenopausal history.
  2. Nonsterile male subjects with sexual partners of childbearing potential must agree to use adequate methods of contraception from CRU admission through Safety Follow-up. Adequate methods of contraception for subjects or partner include the following: condom with spermicidal gel, diaphragm with spermicidal gel, coil (intrauterine device), surgical sterilization, vasectomy, oral contraceptive pill, depo-progesterone injections, progesterone implant (ie, Implanon®), NuvaRing®, Ortho Evra®; if a subject is not sexually active, but becomes active, he or his partner should use medically accepted forms of contraception.
* Body mass index ≥18.0 to ≤34.0 kg/m2, inclusive, at Screening
* Willing to adhere to the prohibitions and restrictions specified in this protocol
* Willing and able to provide written informed consent
* Additionally, for subjects with hepatic impairment:
* Clinical diagnosis of chronic hepatic disease (stable for >3 months) with a documented history of underlying hepatic insufficiency with features of cirrhosis and no acute episodes of illness within 30 days prior to Screening, and no significant change in disease status from Screening to CRU admission (Day -1)
* Hepatic impairment classified as severe using C-P criteria
* A stable medication regimen, defined as not starting new therapy(ies) or significant changing dosage(s) within 30 days prior to dosing on planned Day 1, as determined by the Investigator, Medical Monitor, and/or the Sponsor
* Abnormal laboratory values must be clinically acceptable, as judged by the Investigator, Medical Monitor, and/or the Sponsor.
* Additionally, for healthy matched control subjects with normal hepatic function:
* Each subject will be demographically matched to 1 of the subjects with severe hepatic impairment for sex, age (±10 years), and BMI (±20%).
* No clinically significant illness or disease as determined by medical history, including cardiac, pulmonary, hepatic, biliary, gastrointestinal (GI), endocrinologic, or renal disorders, or cancer within the last 5 years (except localized or in situ cancer of the skin), physical examination, clinical laboratory tests, and 12-lead electrocardiograms (ECGs)
* All laboratory values at Screening and CRU admission fall within normal range or are evaluated as not clinically significant (NCS) by the Investigator if outside normal range. A single test repeat at the discretion of the Investigator is allowed during the Screening Period to determine eligibility.

Exclusion Criteria:

* Presence of clinically significant physical, laboratory, or ECG findings that, in the opinion of the Investigator, Medical Monitor, and/or the Sponsor, may interfere with any aspect of study conduct or interpretation of results including:

  1. Any clinically significant abnormal rhythm
  2. Other ECG abnormalities that are clinically relevant
* Receipt of any investigational agent or study drug within 30 days or 5 half-lives, whichever is longer, prior to CRU admission
* Receipt of any protein- or antibody-based therapeutic agents (eg, growth hormones or monoclonal antibodies) within 3 months prior to dosing on planned Day 1. Note: Influenza vaccine will be allowed if administered >21 days prior to dosing.
* Prior exposure to study drug
* Smoking more than 20 cigarettes (eg, 1 pack) per day or equivalent (eg, e-vapor cigarette, pipe, cigar, chewing tobacco, nicotine patch, nicotine gum); unable or unwilling to refrain from smoking and tobacco use for 2 hours prior to dosing and 4 hours after dose administration.
* History of any serious adverse reaction or hypersensitivity to any inactive component of study drug, unless the reaction is deemed irrelevant to the study by the Investigator, Medical Monitor, and/or the Sponsor
* Existence of any surgical or medical condition that, in the judgment of the Investigator, Medical Monitor, and/or the Sponsor, might interfere with the absorption, distribution, metabolism, or excretion of TE or LP-778902 (including bariatric surgery, cholecystectomy, or any other GI surgery, excepting appendectomy and hernia repair, which are acceptable)
* History of any major surgery within 6 months or anticipated surgery prior to planned CRU admission
* History of renal disease, or significantly abnormal kidney function test (glomerular filtration rate [GFR] <60 mL/min as calculated using the Cockcroft-Gault equation) at CRU admission
* History of any active infection within 30 days prior to Day 1, if deemed clinically significant by the Investigator, Medical Monitor, and/or the Sponsor
* Donation or loss of >500 mL of blood or blood product within 3 months prior to CRU admission
* Women who are breastfeeding or are planning to become pregnant during the study
* Positive serum pregnancy test (females only)
* Positive urine screen for drugs of abuse (not including cotinine) at Screening or CRU admission, unless the result is due to a prescribed medication and is deemed unrelated to the study by the Medical Monitor and/or Sponsor.
* Consumption of alcohol within 3 days hours prior to CRU admission on Day -1 (as confirmed by alcohol breath screen) and for the duration of the confinement period
* Consumption of caffeine- and/or xanthine-containing products (eg, cola, coffee, tea, chocolate) within 72 hours prior to CRU admission (Day -1) and for the duration of the confinement period
* Consumption of grapefruit, Seville oranges, and grapefruit- or Seville orange-containing products within 72 hours prior to CRU admission (Day -1) and for the duration of the confinement period
* Need for special dietary restrictions, unless the restrictions are approved by the Investigator, Medical Monitor, and/or the Sponsor
* Inability or difficulty swallowing whole tablets
* Poor venous access as defined by the Investigator or a designee
* Any other condition that compromises the ability of the subject to provide informed consent or to comply with the objectives and procedures of this protocol, as judged by the Investigator, Medical Monitor, and/or the Sponsor
* Unable or unwilling to cooperate with the Investigator for any reason
* Employee of the Investigator or study center, with direct involvement in the proposed study or other studies under the direction of that Investigator or study center, as well as family members of the employees or the Investigator
* If heparin is to be used during PK sampling, subjects with a history of sensitivity to heparin, or heparin-induced thrombocytopenia, will not be enrolled.
* Administration of gastric acid suppressing agents or short acting octreotide within 30 days or 5 half-lives of the drug, prior to CRU admission
* Use of agents that are known to alter GI motility including, but not limited to, prokinetic agents, antidiarrheals, opiates, antispasmodics, anticholinergics, and antiemetics.
* Additionally, for subjects with hepatic impairment:
* Use of acetaminophen or acetaminophen-containing products within 14 days prior to dosing on planned Day 1 and through Discharge unless deemed acceptable by the Investigator, Medical Monitor, and/or the Sponsor
* Evidence of significant active disease including gastroenterologic (other than hepatic cirrhosis), cardiac (eg, myocardial infarction in the past year, angina, or congestive heart failure), renal, respiratory, endocrine, hematologic, neuropsychiatric, or neoplastic (basal or squamous cell skin cancer is acceptable) disease
* Significant infection or hospitalization within 4 weeks prior to planned Day 1
* Positive for hepatitis B surface antigen (HBsAg; not including hepatitis C virus [HCV] antibody) or positive human immunodeficiency virus (HIV) antibody screens. Note: Subjects with chronic hepatitis C virus (HCV) (duration >6 months) are eligible for enrollment, if stable.
* Primary sclerosing cholangitis or preliminary diagnosed biliary obstruction
* A change in any clinical laboratory value from Screening to Day -1 that is considered by the Investigator, Medical Monitor, and/or the Sponsor to be clinically significant
* History of transplant, portal shunts, recent variceal bleeds, or evidence of hepatorenal syndrome. Note: Creatinine clearance must be ≥60 mL/min using Cockcroft-Gault equation.
* Subjects with a life expectancy less than 3 months
* Additionally, for Healthy Subjects:
* Use of any medications (prescription or over-the-counter), herbal tea, energy drinks, herbal products (eg, St. John's wort, garlic, milk thistle), or supplements/supratherapeutic doses of vitamins within 14 days prior to planned Day 1 and throughout the duration of the study, with the exception of those approved by the Investigator, Medical Monitor, and/or the Sponsor or Sponsor's representative (eg, acetaminophen). Note: The use of typical amounts of garlic used in the preparation of food items is permitted.
* History of hepatic disease, or significantly abnormal liver function tests (>1.5 x upper limit of normal [ULN]) at Screening. Note: Isolated bilirubin >1.5 x ULN is acceptable if bilirubin is fractionated and direct bilirubin is <35%.
* Positive hepatitis panel (including HBsAg and HCV antibody) or positive HIV antibody screens
* History of any clinically relevant psychiatric, renal, hepatic, pancreatic, endocrinologic, cardiovascular, neurological, hematological
* History of alcohol or substance abuse within 2 years prior to Screening per Diagnostic and Statistical Manual of Mental Disorders, 5th Edition criteria
* Concurrent conditions that could interfere with safety and/or tolerability measurements

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2017-11-28 (Actual); Primary Completion 2018-06-15 (Actual); Study Completion 2018-06-15 (Actual)

PRIMARY OUTCOMES:
Maximum observed concentration of telotristat ethyl | 4 days
Time of maximum observed concentration of telotristat ethyl | 4 days
Area under the plasma concentration-time curve beginning from the first dose until the last quantifiable concentration of telotristat ethyl | 4 days

SECONDARY OUTCOMES:
Number of adverse events | Up to 9 days

CONTACTS AND LOCATIONS:
Overall Officials: Suman Wason, MD, Study Director — Lexicon Pharmaceuticals, Inc.
Locations (3):
- United States (3):
  - Lexicon Investigational Site, Miami, Florida
  - Lexicon Investigational Site, Orlando, Florida
  - Lexicon Investigational Site, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: Undecided